CLINICAL TRIAL: NCT01050504
Title: Molecular Correlates of Sensitivity and Resistance to Therapy in Genitourinary Malignancy
Brief Title: Collecting and Studying Blood and Tissue Samples From Patients With Locally Recurrent or Metastatic Prostate or Bladder/Urothelial Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6932; NCI-2014-01087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6932p; 6932 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1712006 (Other: Fred Hutch/University of Washington Cancer Consortium); P50CA097186 (NIH)
Record Dates: First submitted 2009-09-30; First posted 2010-01-15 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Localized Renal Pelvis and Ureter Urothelial Carcinoma; Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Soft Tissues; Metastatic Renal Pelvis and Ureter Urothelial Carcinoma; Recurrent Bladder Carcinoma; Recurrent Prostate Carcinoma; Recurrent Renal Pelvis and Ureter Urothelial Carcinoma; Stage IV Bladder Cancer AJCC v7; Stage IV Bladder Urothelial Carcinoma AJCC v7; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-correlative (blood and tissue collection): Patients undergo collection of blood and tissue samples for analysis via mutation mapping, DNA sequencing, gene expression microarray, and gene profiling.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This study collects and studies tissue and blood samples from patients with prostate or bladder/urothelial cancer that has recurred (come back) at or near the same place as the original (primary) tumor or has spread to other parts of the body. Studying samples of blood and tissue samples from patients with prostate or bladder/urothelial cancer in the laboratory may help doctors learn more about new biomarkers, potential drug targets, and resistance developing in response to treatment. It may also help doctors find better ways to treat the cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo collection of blood and tissue samples for analysis via mutation mapping, DNA sequencing, gene expression microarray, and gene profiling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized and/or metastatic bladder/urothelial or prostate cancer who have disease in the primary organ, biopsy accessible bone metastases (collaborating radiologists will determine if bone metastasis is appropriate for biopsy) or soft tissue metastases are eligible; men and women without cancer are eligible to have blood or normal tissue collected if acquired as part of non-research procedures (e.g. transurethral resection of the prostate or bladder); in patients without malignancy, no additional tissue beyond that necessary for care will be procured
* Ability to adequately understand and give informed consent
* Local or metastatic disease to soft tissue or bone at sites accessible to biopsy with minimal risk of complications Or the ability to obtain tissue with minimal risk of complication from a surgical procedure being conducted as a part of another research study Or for standard of care purposes or patients who have archival tissue collected for research or standard of care who are willing to donate archival tissue for this study
* Alternatively, men and women without cancer or who are at risk of developing cancer are eligible to have blood or normal tissue collected if acquired; tissue will only be acquired as part of non-research procedures (e.g. transurethral resection of the prostate or bladder; in patients without malignancy, no additional tissue beyond that necessary for care will be procured
* Platelet count > 50,000
* White blood cell (WBC) > 1,500
* Hemoglobin (Hgb) > 8.0
* International normalized ratio (INR) < 1.5
* Partial thromboplastin time (PTT) < 45
* No history of excessive unexplained bleeding from previous surgery

Exclusion Criteria:

* Patients unable to stop chronic anticoagulation with warfarin or Lovenox for less than 3 days
* Serious or uncontrolled infection
* Treatment with a vascular endothelial growth factor (VEGF) inhibitor (such as Avastin) within the past 28 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with prostate or bladder/urothelial cancer treated in genitourinary oncology practices at University of Washington Medical Center, Seattle Cancer care Alliance and Harborview Medical Center and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-08; Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
DNA genomic sequencing | Up to 6 years
Gene expression profile using microarray assays | Up to 6 years
Mutation mapping using the OncoMap and other genotyping techniques | Up to 6 years

SECONDARY OUTCOMES:
Expression of androgen metabolic enzymes by quantitative real time-polymerase chain reaction | Up to 6 years
Proteomic profile | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Montgomery, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No